CLINICAL TRIAL: NCT04662866
Title: Glucose Metabolism in South Asian Women With IGT or IFG. DIAbetes in South Asians - DIASA 3: A 12-week Intervention Trial With Oral Antidiabetic Medication to Improve Hepatic and Whole Body Insulin Sensitivity
Brief Title: Effects of Glucose Lowering Agents in South Asian Women With Impaired Glucose Tolerance or Impaired Fasting Glucose
Acronym: DIASA3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Norwegian Diabetes Association (Other); South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); University of Glasgow (Other)
Responsible Party: Principal Investigator, Kåre Inge Birkeland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24993
Record Dates: First submitted 2020-11-16; First posted 2020-12-10 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Impaired Glucose Tolerance; Insulin Sensitivity; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Glucose Metabolism Disorders | interventions — Metformin; Biguanides; Thiazolidinediones

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (RCT), 4 parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin (Active Comparator): Metformin 500 mg x 1, morning, for 2 weeks, then Metformin 500 mg x 2, morning and evening for 10 weeks.
  Interventions: Drug: Metformin capsule 500 mg, Empagliflozin encapsulated tablet 10 mg, Pioglitazone encapsulated tablet 30 mg, Linagliptin encapsulated tablet 5 mg
- Empagliflozin (Active Comparator): Empagliflozin 10 mg x 1, morning, for 2 weeks, then Empagliflozin 10 mg morning + Placebo evening for 10 weeks.
  Interventions: Drug: Metformin capsule 500 mg, Empagliflozin encapsulated tablet 10 mg, Pioglitazone encapsulated tablet 30 mg, Linagliptin encapsulated tablet 5 mg
- Linagliptin (Active Comparator): Linagliptin 5 mg x 1, morning, for 2 weeks, then Linagliptin 5 mg morning + Placebo evening for 10 weeks.
  Interventions: Drug: Metformin capsule 500 mg, Empagliflozin encapsulated tablet 10 mg, Pioglitazone encapsulated tablet 30 mg, Linagliptin encapsulated tablet 5 mg
- Pioglitazone (Active Comparator): Pioglitazone 30 mg x 1, morning, for 2 weeks, then Pioglitazone 30 mg morning + Placebo evening for 10 weeks.
  Interventions: Drug: Metformin capsule 500 mg, Empagliflozin encapsulated tablet 10 mg, Pioglitazone encapsulated tablet 30 mg, Linagliptin encapsulated tablet 5 mg

INTERVENTIONS:
Drug: Metformin capsule 500 mg, Empagliflozin encapsulated tablet 10 mg, Pioglitazone encapsulated tablet 30 mg, Linagliptin encapsulated tablet 5 mg — Comparison of 4 different antihyperglycemic drugs
  Other Names: biguanide, glitazone, sodium glucose transport inhibitor, dipeptidyl peptidase inhibitor

SUMMARY:
This study will test the effect of four common oral anti-diabetic agents on hepatic insulin sensitivity in South Asian women with impaired glucose tolerance or impaired fasting glucose. In a 12-week, double-blind, randomized controlled intervention trial, the following drugs will be tested head-to-head: Metformin, Pioglitazone, Empagliflozin and Linagliptin. Additional, exploratory outcomes include whole body insulin sensitivity, insulin secretion and other markers of glucose and lipid metabolism, measured by the euglycemic clamp with stable isotope tracer dilution, indirect calorimetry and CT-measurements of abdominal adipose tissue compartment volumes and hepatic and pancreatic volume and attenuation.

The study is part of the DIASA - DIAbetes in South Asians - Research Programme, which aims to find ways to improve both prevention and treatment of type 2 diabetes in people of South Asian ethnicity.

DETAILED DESCRIPTION:
Background: South Asians (SA) have a high prevalence of type 2 diabetes (T2D). SA i Norway develop T2D approximately 10 years earlier than Nordic subjects (NO).T2D in SA is often poorly regulated with increased risk of complications.

Research hypothesis: South Asian subjects with Impaired glucose tolerance (IGT) or impaired fasting glucose (IFG) have a high degree of hepatic insulin resistance. Treatment with certain oral antidiabetic drugs will improve hepatic insulin sensitivity more than others.

Primary objective: To assess which of four oral antidiabetic medications is most effective in improving hepatic insulin sensitivity in women of South Asian origin with IFG/IGT.

Study design: Single-center, randomized, double-blind intervention trial with 4 parallel treatment arms: 1) Metformin 2) Pioglitazone 3) Empagliflozin 4) Linagliptin.

Endogenous glucose production (EGP) and hepatic and whole body insulin sensitivity will be assessed by a 2-step euglycemic, hyperinsulinemic clamp with deuterated glucose tracer. In addition, glucose and lipid metabolism will be assessed by indirect calorimetry (IC), insulin secretion by an oral glucose tolerance test (OGTT), and fatty infiltration in liver by computer tomography (CT).

Recruitment: From South Asian women with IFG/IGT who participated in DIASA 1.

Duration of study: 14 weeks, with a total of four study visits, every 4 weeks, plus two CT scans, at baseline and 12 weeks, and one end of study follow-up telephone visit at 14 weeks. The project is expected to last a maximum of 3 years.

Study population: Women ≥ 18 years of age of South Asian ethnicity with IGT/IFG.

Criteria for evaluation: Efficacy outcome will include evaluation of change in EGP from baseline to 12 weeks. Laboratory parameters of glucose and lipid metabolism. Questionnaires with physical activity and food frequency. Safety and tolerability will be assessed by clinical adverse events and laboratory measurements from randomization to 14 weeks.

Primary outcome: Difference between treatment arms in change in EGP from baseline to 12 weeks.

Explorative outcomes: Difference between treatment arms in change from randomisation to 12 weeks in:

* whole body insulin sensitivity
* HbA1c
* glucose and lipid metabolism measured by IC
* fatty infiltration in liver and visceral adipose tissue.

Statistical Methods: One-way ANOVA, Multiple regression analyses, Paired samples t-tests, longitudinal analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give informed consent
2. Woman ≥ 18 years of age
3. Of South Asian origin
4. Participated in the DIASA 1 study (i.e. has had previous gestational diabetes (GDM) in last pregnancy). A period of 3 months after the 3-year limit since childbirth after GDM is seen as acceptable for inclusion.
5. Impaired glucose tolerance (2-hour glucose value ≥7.8 and < 11.1 mmol/l) and/or impaired fasting glucose (fasting plasma glucose ≥ 6.1 and < 7.0 mmol/l) diagnosed in DIASA 1

Exclusion Criteria:

1. Known type 2 diabetes
2. Known type 1 diabetes
3. Fasting or 2-hour glucose values outside the inclusion criteria if the subject according to protocol needs to undergo an OGTT at baseline in DIASA 3
4. Pregnant or fully lactating at randomisation or planned during study period.
5. Not willing to practice a highly effective birth control method* prior to initial dose, during study and for 2 weeks after the last administration of study drug.
6. Concomitant use of any antidiabetic medication
7. Concomitant use of fibrates or rifampicin
8. Radiological examinations iodine containing contrast the previous week before randomisation, or planned during the study period.
9. Known serious illness such as cancer (except in situ carcinoma) during past 5 years.
10. Previous radiation therapy directed towards the pelvic area.
11. Heart failure New York Heart Association (NYHA) class I-IV.
12. Estimated glomerulus filtration rate (eGFR) < 60 ml/min/1,73m2
13. Chronic liver disease with serum levels of aspartate aminotransferase (ASAT) or alanine amino transferase (ALAT) > 5 x upper limit of normal (ULN) or known impaired liver function (INR > 1.5, Albumin < 20 g/l, Bilirubin > 20 g/l.
14. Active infectious disease at inclusion
15. Use of systemic corticosteroids > 14 days within last 3 months before inclusion
16. Hypothyroidism where substitution with levothyroxine has not been stable for the last 3 months or with thyroid stimulating hormone (TSH) outside normal limits.
17. A history of bullous pemphigoid
18. A history of acute or chronic pancreatitis
19. Previous or present acute metabolic acidosis.
20. Known hypersensitivity to any of the active ingredients or additives in the study medication or placebo capsules.
21. Macroscopic haematuria not previously examined
22. History of major surgical procedures within 3 months prior to inclusion or planned during study period.
23. Any condition which in the investigator's opinion would jeopardize the subject's safety or compliance with the protocol.

    * Birth control methods which may be considered as highly effective: Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system ( IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Endogenous glucose production during fasting | After 12 weeks on respective drugs
  Difference between treatment arms in change from baseline to 12 weeks in endogenous glucose production during fasting measured by the deuterated glucose tracer dilution method in umol/(kg fat free mass x minutes)

OTHER OUTCOMES:
Endogenous glucose production during hyperinsulinemia | After 12 weeks on respective drugs
  Difference between treatment arms in change from baseline to 12 weeks in endogenous glucose production measured by the deuterated glucose tracer dilution method during euglycaemic clamp in umol/(kg fat free mass x minutes)
Whole body insulin sensitivity | After 12 weeks on respective drugs
  Difference between treatment arms in change from baseline to 12 weeks in whole body insulin sensitivity measured by euglycemic clamp derived total glucose disposal in umol/(kg fat free mass x minutes)
Insulin secretion | After 12 weeks on respective drugs
  Difference between treatment arms in change in insulin secretion from baseline to 12 weeks, measured by the insulinogenic index, i.e. the change in serum insulin (pmol/l) from 0 to 30 min divided by the change in plasma glucose (mmol/l) from 0 to 30 minutes of an oral glucose tolerance test.
Liver fat | After 12 weeks on respective drugs
  Explore the difference between treatment arms in change in fatty infiltration in the liver measured as the attenuation in CT-measured regions of interest from baseline to 12 weeks.
Glycemia | After 12 weeks on respective drugs
  Difference between treatment arms in change in HbA1c in mmol/mol from baseline to 12 weeks .
Pancreatic fat | After 12 weeks on respective drugs
  Explore the difference between treatment arms in change in fatty infiltration of the pancreas measured as the attenuation in CT-measured regions of interest
Intraabdominal fat | After 12 weeks on respective drugs
  Explore the difference between treatment arms in change in visceral fat volume, in cubic centimeters, from baseline to 12 weeks, on abdominal CT scans running from the top of the diaphragm to the iliac crest.

CONTACTS AND LOCATIONS:
Overall Officials: Kåre I Birkeland, MD, PhD, Principal Investigator — Professor
Locations (1):
- Oslo University Hospital, Aker Hospital, Oslo, Norway